CLINICAL TRIAL: NCT01482325
Title: SNIPE:SuperSTAT 2.0 Noninvasive Blood Pressure Algorithm Enhancement
Brief Title: SuperSTAT 2.0 Noninvasive Blood Pressure Algorithm Enhancement
Acronym: SNIPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The business decided not to pursue the study at this time.
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 118.02-2011-GES-0002
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Blood Pressure (Low, Normal, High)
MeSH Terms: interventions — Blood Pressure Monitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects requiring blood pressure monitoring (Experimental): Any subject (neonate-adult) requiring hospital or clinic blood pressure monitoring
  Interventions: Device: Blood pressure monitoring with GE Healthcare DASH2500 Patient Monitor

INTERVENTIONS:
Device: Blood pressure monitoring with GE Healthcare DASH2500 Patient Monitor — 10-20 Non-Invasive Blood Pressure readings on investigational software in the DASH2500 Patient Monitor

SUMMARY:
The primary objective of this study is to show that the noninvasive blood pressure software algorithm meets engineering requirements.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent or have a legally authorized representative including a parent or guardian provide written informed consent
* Ability of a minor subject ages 7 to 18 to provide written assent
* Ability to have multiple noninvasive blood pressures taken at one sitting
* Ability to apply three lead ECG, if needed for investigation
* Ability to detect the natural presence of an irregular pulse, for irregular pulse studies

Exclusion Criteria:

* Any subject who cannot tolerate multiple blood pressure measurements
* Any subject who cannot undergo 3-lead ECG, if needed
* Any subject deemed unstable by the principal investigator
* Any subject for whom precautions are necessary because of communicable disease
* Any subject that has a known disease or condition compromises musculoskeletal integrity
* Any subject that has a known disease or condition that contraindicates use of an NIBP cuff and ECG patches on the skin.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - St. Josephs Hospital, Milwaukee, Wisconsin
  - Wisconsin Heart Hospital, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Requiring Blood Pressure Monitoring: St. Joseph's Hospital (001), there were 21 subjects screened, of which five were screen failures and 16 subjects completed the study. Wisconsin Heart Hospital (002), there were 25 subjects screened, of which 10 were screen failures and 15 subjects completed the study.
  There were enrollment criteria followed by both Site 001 and Site 002 that were provided by the study's GEHC engineer in order to test the SuperSTAT algorithm. Each set of subjects enrolled under the required enrollment criteria were tested by the GEHC engineer.
Period: Overall Study
Arm/Group | Subjects Requiring Blood Pressure Monitoring
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No analysis was performed, study prematurely terminated.
Arm/Group | Subjects Requiring Blood Pressure Monitoring
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.49 (32.74)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 18
    Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Data Collection for Engineering Development
Description: This was a data collection for engineering development to demonstrate SuperSTAT 2.0 NIBP software algorithm meets the engineering specifications. Engineers reviewed data produced by each blood pressure determination to work on new software algorithm in development. This was not conducted as program was terminated prematurely.
  Software iterations are not pre-defined.
Time Frame: After each iteration of software development
Population: Subject analysis was not performed because study was prematurely terminated. Work on the project ceased when it was terminated.The study was intended to have the engineers review data produced by each blood pressure determination to work on new software algorithm in development. This was not and will not be conducted.
Arm/Group | Subjects Requiring Blood Pressure Monitoring
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Subjects Requiring Blood Pressure Monitoring: Any subject (neonate-adult) requiring hospital or clinic blood pressure monitoring
  Blood pressure monitoring with GE Healthcare DASH2500 Patient Monitor: 10-20 Non-Invasive Blood Pressure readings on investigational software in the DASH2500 Patient Monitor
  At Site #001 - St. Joseph's Hospital, there were 21 subjects screened, of which five were screen failures and 16 subjects completed the study. There were no adverse events reported.
  At Site #002 - Wisconsin Heart Hospital, there were 25 subjects screened, of which 10 were screen failures and 15 subjects completed the study. There were no adverse events reported.
Arm/Group | Subjects Requiring Blood Pressure Monitoring
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No